CLINICAL TRIAL: NCT06249477
Title: Weight Loss and Physical Activity Lifestyle Interventions In Post Liver And Kidney Transplants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Society of Transplantation (Unknown)
Responsible Party: Principal Investigator, Leigh Anne Dageforde, Assistant Professor of Surgery, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021P003412
Record Dates: First submitted 2024-01-22; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Weight Loss; Lifestyle Factors
Keywords: Transplant; Weight loss; Lifestyle intervention; Obesity management
MeSH Terms: conditions — Weight Loss | interventions — Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Patients receive a wrist activity monitor and a scale. They are also followed with monthly calls ensuring adequate functioning of devices and receiving case-specific nutritional guidance.
  Interventions: Device: Wrist activity tracker and scale
- Group intervention group (Experimental): In addition to receiving a wrist activity monitor, scale, and being followed with monthly calls, patients in this arm received every other month nutritional coaching group sessions on topics related to nutrition and physical activity to promote education and lifestyle changes
  Interventions: Device: Wrist activity tracker and scale; Behavioral: Nutritional Coaching group sessions

INTERVENTIONS:
Device: Wrist activity tracker and scale — Wrist activity tracker used to evaluate number of steps, heart rate, and frequency of usage of the devices to monitor activity. Scale used to record a patient's weight value.
  Other Names: Fitbit Charge 4
Behavioral: Nutritional Coaching group sessions — Nutritional coaching group sessions held via zoom and performed by a certified clinical nutritionist regarding nutrition, and physical activity specific for weight loss.
  Arms: Group intervention group

SUMMARY:
This research project seeks to learn more about how lifestyle interventions can help liver and kidney transplant recipients achieve weight loss goals. The investigators want to evaluate if an intervention using weight and activity wrist monitors, as well as nutritional coaching group sessions is acceptable and useful for post-transplant patients aiming for weight loss. All participants will be given a wrist activity monitor, and a scale. Half of participants will be invited to participate in the nutritional coaching group sessions. The research team will look at weight loss, devices' usage, and satisfaction, and see if there are any difference among the two groups.

DETAILED DESCRIPTION:
This project aims to understand feasibility, acceptability, and appropriateness of using connected health services (use of Fitbit and Scale), and nutritional coaching group sessions as a lifestyle intervention for post-transplant patients seeking weight loss. Secondarily, the investigators aim to assess effectiveness of the intervention to generate weight loss. Enrolled patients will receive a wrist activity tracker (Fitbit Charge 4) and a scale, of which information synchronizes to the electronic health record. Steps, usage, and weight values will be recorded and analyzed from the devices. All patients will be followed with monthly calls to assess issues with devices, and address case-specific questions. Simultaneously, half of the patients will be randomized to receive every other month nutritional coaching group sessions on topics related to nutrition and physical activity. Patients will have an in-person follow-up appointment where laboratory values, body measurements, and physical and mental readiness for weight loss surveys and scales will be applied at 6 and 12-months. Patients that don't accomplish weight loss goal at 6 months will be invited to cross over to the nutritional coaching group sessions intervention arm.

ELIGIBILITY:
Inclusion Criteria:

* Prior liver or kidney transplant recipient
* BMI >=30
* 6 months to 10 years post-transplant
* Stable immunosuppression as defined by no treatment for rejection in the past 3 months
* Access to Smartphone or computer
* Able to provide informed consent

Exclusion Criteria:

* Dual and/or simultaneous organ kidney and liver transplant
* Any type of other prior transplant
* Age <= 18 years old
* Treatment for rejection within the last 3 months
* Major infection requiring hospitalization within the last 3 months
* Relisting for liver transplant or returned to dialysis for kidney transplant
* Physical inability to participate in lifestyle intervention activity recommendations
* Patients that are actively enrolled in a weight center program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention | 12 months (All study duration)
  The Feasibility of Intervention Measurement (FIM) is a previously-validated survey tool used in implementation science, and answered by participants, that uses a Likert scale from 1 to 5 to evaluate feasibility of the proposed intervention. A score greater than or equal to 4 is considered acceptable feasibility.
Acceptability of intervention | 12 months (All study duration)
  The Acceptability of Intervention Measurement (AIM) is a previously-validated survey tool used in implementation science, and answered by participants, that uses a Likert scale from 1 to 5 to evaluate acceptability of the proposed intervention. A score greater than or equal to 4 is considered adequate acceptability.
Rate of highly satisfied Patients | 12 months (All study duration)
  Patient-completed satisfaction questionnaires will be evaluated using a Likert scale from 1 to 5 with five being very satisfied and one being very unsatisfied. Satisfaction surveys were asked separately for the use of devices (Fitbit and smart scale), every other month follow-up calls, and every other month group sessions. An additional overall satisfaction score was also obtained for the entire intervention. High satisfaction will be considered the proportion of "somewhat satisfied" and "very satisfied" answers.
Wrist activity tracker usage rate | 12 months (All study duration)
  Usage rate will be calculated as the proportion of days in which steps are logged in relation to the number of days per month.

SECONDARY OUTCOMES:
Weight change percentage | 12 months (All study duration)
  Target Weight change percentage will be considered a greater than or equal to 2.5% loss at 6 months, and greater than or equal to 5% weight loss over the course of the 12-month period.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh A Dageforde, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data available to other researchers since all data analysis and publications that derive from the information collected through this trial will be handled and analyzed by the current research team. No additional analyses or data management other than the originally intended is planned or allowed.

REFERENCES:
- [Background] Estes C, Razavi H, Loomba R, Younossi Z, Sanyal AJ. Modeling the epidemic of nonalcoholic fatty liver disease demonstrates an exponential increase in burden of disease. Hepatology. 2018 Jan;67(1):123-133. doi: 10.1002/hep.29466. Epub 2017 Dec 1. PMID 28802062
- [Background] Saeed N, Glass L, Sharma P, Shannon C, Sonnenday CJ, Tincopa MA. Incidence and Risks for Nonalcoholic Fatty Liver Disease and Steatohepatitis Post-liver Transplant: Systematic Review and Meta-analysis. Transplantation. 2019 Nov;103(11):e345-e354. doi: 10.1097/TP.0000000000002916. PMID 31415032
- [Background] Germani G, Laryea M, Rubbia-Brandt L, Egawa H, Burra P, O'Grady J, Watt KD. Management of Recurrent and De Novo NAFLD/NASH After Liver Transplantation. Transplantation. 2019 Jan;103(1):57-67. doi: 10.1097/TP.0000000000002485. PMID 30335694
- [Background] Wang X, Li J, Riaz DR, Shi G, Liu C, Dai Y. Outcomes of liver transplantation for nonalcoholic steatohepatitis: a systematic review and meta-analysis. Clin Gastroenterol Hepatol. 2014 Mar;12(3):394-402.e1. doi: 10.1016/j.cgh.2013.09.023. Epub 2013 Sep 25. PMID 24076414
- [Background] Cotter TG, Charlton M. Nonalcoholic Steatohepatitis After Liver Transplantation. Liver Transpl. 2020 Jan;26(1):141-159. doi: 10.1002/lt.25657. Epub 2019 Nov 25. PMID 31610081
- [Background] Wadden TA, Brownell KD, Foster GD. Obesity: responding to the global epidemic. J Consult Clin Psychol. 2002 Jun;70(3):510-25. doi: 10.1037//0022-006x.70.3.510. PMID 12090366
- [Background] O'Brien T, Russell CL, Tan A, Mion L, Rose K, Focht B, Daloul R, Hathaway D. A Pilot Randomized Controlled Trial Using SystemCHANGE Approach to Increase Physical Activity in Older Kidney Transplant Recipients. Prog Transplant. 2020 Dec;30(4):306-314. doi: 10.1177/1526924820958148. Epub 2020 Sep 10. PMID 32912051
- [Background] Neale J, Smith AC. Cardiovascular risk factors following renal transplant. World J Transplant. 2015 Dec 24;5(4):183-95. doi: 10.5500/wjt.v5.i4.183. PMID 26722646
- [Background] Chen G, Gao L, Li X. Effects of exercise training on cardiovascular risk factors in kidney transplant recipients: a systematic review and meta-analysis. Ren Fail. 2019 Nov;41(1):408-418. doi: 10.1080/0886022X.2019.1611602. PMID 31106657
- [Background] Andres A, Saldana C, Gomez-Benito J. The transtheoretical model in weight management: validation of the processes of change questionnaire. Obes Facts. 2011;4(6):433-42. doi: 10.1159/000335135. Epub 2011 Nov 25. PMID 22248993
- [Background] Andres A, Saldana C, Gomez-Benito J. Establishing the stages and processes of change for weight loss by consensus of experts. Obesity (Silver Spring). 2009 Sep;17(9):1717-23. doi: 10.1038/oby.2009.100. Epub 2009 Apr 9. PMID 19360014
- [Background] Steinberg DM, Bennett GG, Askew S, Tate DF. Weighing every day matters: daily weighing improves weight loss and adoption of weight control behaviors. J Acad Nutr Diet. 2015 Apr;115(4):511-8. doi: 10.1016/j.jand.2014.12.011. Epub 2015 Feb 12. PMID 25683820
- [Background] Palmeira AL, Teixeira PJ, Branco TL, Martins SS, Minderico CS, Barata JT, Serpa SO, Sardinha LB. Predicting short-term weight loss using four leading health behavior change theories. Int J Behav Nutr Phys Act. 2007 Apr 20;4:14. doi: 10.1186/1479-5868-4-14. PMID 17448248
- [Background] Takacs J, Pollock CL, Guenther JR, Bahar M, Napier C, Hunt MA. Validation of the Fitbit One activity monitor device during treadmill walking. J Sci Med Sport. 2014 Sep;17(5):496-500. doi: 10.1016/j.jsams.2013.10.241. Epub 2013 Oct 31. PMID 24268570
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- See also: World Health Organization [WHO]. (2014). Obesity and Overweight. Fact Sheet N 311, Geneva: World Health Organization. — https://www.who.int/news-room/fact-sheets/detail/obesity-and-overweight